CLINICAL TRIAL: NCT01818570
Title: A Single-center, Randomized, Double-blind, Cross-over Trial in Healthy Volunteers Investigating the Local Efficacy and Safety of a Single Intra-luminal Administration of PPC-5650 on Reflux Pain and Hyperalgesia During Multimodal Stimulation of the Esophagus
Brief Title: A Study of Local Effect and Safety of a Single PPC-5650 Dose on Reflux Pain During Pain Stimulation in the Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROS-002
Record Dates: First submitted 2013-03-22; First posted 2013-03-26 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Gastroesophageal Reflux; Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo solution (Placebo Comparator): A 100 ml placebo solution will be administered through an esophageal probe. 100 ml will be administered as an infusion with a rate of 7ml/min. Healthy volunteers will be treated with placebo in one out of three visit days.
  Interventions: Drug: Placebo
- PPC-5650 (Active Comparator): PPC-5650 is a "asic-sensing ion channel"-1a antagonist that can block the acid-sensing ion channels, leading to a reduction in the pain signal under up-regulated conditions. A dose of 2.5 mg PPC-5650 in a 100 ml solution will be administered through an esophageal probe to assess local effects. 100 ml will be administered as an infusion with a rate of 7ml/min. Healthy volunteers will be treated with PPC-5650 in one out of three visit days.
  Interventions: Drug: PPC-5650

INTERVENTIONS:
Drug: PPC-5650 — A dose of 2.5 mg PPC-5650 in a 100 ml solution will be administered to the esophagus with an infusion rate of 7ml/min in one out of three visit days.
  Arms: PPC-5650
Drug: Placebo — A 100 ml placebo solution will be administered to the esophagus with an infusion rate of 7ml/min in one out of three visit days.
  Arms: Placebo solution

SUMMARY:
The purpose of this trial is to evaluate the effect of a single PPC-5650 dose in a human pain model including multimodal (mechanical, thermal, electrical, chemical) stimulations of the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study specific procedures
* Able to read and understand Danish.
* Healthy i.e. no history of chronic or recurrent pain rewarding diseases
* Able to co-operate and tolerate the experimental procedures (as assessed in the training visit)
* No over the counter medication 24h before the three visits
* No medications in the study period
* BMI 18.5-35.0
* Caucasian
* No symptoms of Gastroesophageal reflux disease
* All men must use a safe method of contraception during the study period

Exclusion Criteria:

* Any clinically relevant abnormal values from the laboratory tests on hematology, clinical chemistry, and/or urine analyses, as judged by the investigator.
* Participation in any other clinical trial within three months prior to the training day.
* Alcohol or drug abuse.
* Mental illnesses
* Allergic to the active ingredient in the investigational medicinal product

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain scores recorded after multimodal pain stimulations (mechanical, thermal, electrical, and chemical) | 4 hours

SECONDARY OUTCOMES:
Number of observed adverse effects (safety profile) and changes in size of referred pain area | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, Professor, Principal Investigator — Mech-Sense, Department of Medical Gastroenterology, Aalborg Hospital
Locations (1):
- Mech-Sense, Department of Medical Gastroenterology, Aalborg University Hospital, Aalborg, Jutland, Denmark

REFERENCES:
- [Derived] Olesen AE, Nielsen LM, Larsen IM, Drewes AM. Randomized clinical trial: efficacy and safety of PPC-5650 on experimental esophageal pain and hyperalgesia in healthy volunteers. Scand J Gastroenterol. 2015 Feb;50(2):138-44. doi: 10.3109/00365521.2014.966319. Epub 2014 Dec 8. PMID 25483563